CLINICAL TRIAL: NCT02496065
Title: A Phase 1 Exploratory Study of the Safety and ex Vivo Fluorescence of BLZ-100 Administered by Intravenous Injection in Adult Subjects With Solid Tumors Undergoing Surgery
Brief Title: Exploratory Study of Safety and ex Vivo Fluorescence of BLZ-100 in Adult Subjects With Solid Tumors Undergoing Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Blaze Bioscience Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BB-005
Record Dates: First submitted 2015-07-08; First posted 2015-07-14 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Tumors, Breast
Keywords: breast cancer; BLZ-100; Tumor Paint; breast tumors
MeSH Terms: conditions — Breast Neoplasms | interventions — tozuleristide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BLZ-100 (Experimental)
  Interventions: Drug: BLZ-100

INTERVENTIONS:
Drug: BLZ-100
  Other Names: Tumor Paint

SUMMARY:
Surgery is the primary treatment modality for many types of cancer and the extent of surgical resection is directly related to patient survival. However, it is often difficult for surgeons to distinguish normal from neoplastic tissue or to detect metastatic disease or tumor-infiltrated lymph nodes. In some sites, surgical precision is also required to avoid damage to critical normal tissues. The purpose of this exploratory study is to evaluate the intra-operative and ex vivo fluorescence of BLZ-100 in tumor samples from subjects with breast cancer.

DETAILED DESCRIPTION:
Subjects diagnosed to have breast cancer for which surgical resection is clinically indicated will be enrolled in this study.

Upon obtaining signed informed consent, subjects will enter a Screening Period for up to 14 days to determine eligibility. Subjects meeting all of the inclusion and none of the exclusion criteria will be eligible to participate in the study.

All subjects entered into the study will be required to arrive at the hospital (or Phase 1 unit if applicable) for BLZ-100 administration at least 2 hours before their scheduled surgical procedure. Following administration of BLZ-100, subjects will be continuously monitored for safety and any allergic reaction occurrence for 30 minutes; thereafter, subjects will be evaluated for 7 days after drug administration. All subjects will be followed for at least 30 days following drug administration to monitor for SAEs.

Tumor samples will be imaged in situ and ex vivo with the SIRIS imaging system or equivalent device, processed, and sent to a central laboratory to be evaluated for ex vivo fluorescence using the Odyssey® CLx imaging system.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject aged 18 years or older.
2. Diagnosed solid tumor scheduled for surgical excision. Subjects with recurrent disease will be eligible only if the duration between last tumor surgery and scheduled new surgery is ≥3 months.
3. Able to provide written informed consent.
4. If of child-bearing potential, agree to continued use of two reliable methods of contraceptive from study entry (time of informed consent) through 30 days after BLZ-100 administration. Male subjects with vasectomy do not need to use a second form of contraceptive.
5. Available for all study visits and able to comply with all study requirements.

Exclusion Criteria:

1. Suspected central nervous system (CNS) tumor(s) or sarcoma.
2. Female who is lactating/breastfeeding.
3. Female with a positive pregnancy test or who is planning to become pregnant during the duration of the study.
4. Karnofsky Performance Status of <60%.
5. Any of the following laboratory abnormalities at Screening:

   1. Neutrophil count <1.5 x 109/L
   2. Platelets <75 x 109/L
   3. Hemoglobin <10 g/dL (may be determined following transfusion)
   4. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 x upper limit of normal (ULN)
   5. Total bilirubin >1.5 x ULN (unless Gilbert's syndrome or extrahepatic source as denoted by increased indirect bilirubin fraction)
   6. International Normalized Ratio (INR) >1.5 x ULN
   7. Creatinine >1.5 x ULN
6. QTc prolongation >480 msec.
7. History of hypersensitivity or allergic reactions requiring corticosteroids, epinephrine, and/or hospitalization.
8. Uncontrolled asthma or asthma requiring oral corticosteroids.
9. Known or suspected sensitivity to diagnostic imaging contrast agents.
10. Known or suspected sensitivity to indocyanine green (ICG).
11. Unstable angina, myocardial infarction, known or suspected transient ischemic events, or stroke within 24 weeks of start of Screening.
12. Uncontrolled hypertension.
13. Initiation of new photosensitizing drugs within 30 days of Screening.
14. Use of any ongoing medications which might generate fluorescence or, according to the medication label, might generate a photochemical reaction. These include haematoporphyrin derivatives and purified fractions, Photofrin®, and the precursors of protoporphyrin IX (5-Aminolevulinic acid) used in Gliolan or Hexvix.
15. Receipt of an investigational drug or device within 30 days of enrollment.
16. Prior treatment with BLZ-100.
17. Any concurrent condition, including psychological and social situations, which, in the opinion of the investigator, would adversely impact the subject or the interpretation of the study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Seven days after study drug administration
  Safety will be assessed by physical examination and measurement of vital signs and laboratory safety parameters. These assessments will be used to determine whether a subject experienced an AE.

SECONDARY OUTCOMES:
Fluorescent signal from excised tumor surgical specimens | Post-tumor excision (approximately 2 hours post BLZ-100 dosing)
  Ex vivo fluorescence of excised tumor specimens will be evaluated with the SIRIS or equivalent imaging device and Odyssey imaging system.
Change of concentration of BLZ-100 in the blood | 5, 15, and 30 minutes post BLZ-100 administration
  BLZ-100 levels in blood will be analyzed by chemical means and these data will be used to calculate pharmacokinetic parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Kristi M Harrington, MD, Principal Investigator — Overlake Medical Center, Overlake Medical Clinics
Locations (2):
- United States (2):
  - Overlake Medical Center, Bellevue, Washington
  - University of Washington Medical Center, Seattle, Washington